CLINICAL TRIAL: NCT04008615
Title: Comparison of the Cardiopulmonary and Gaz-exchange Response Between the Six-minute Stepper Test and the Incremental Cardiopulmonary Exercise Testing in Patients With Chronicle Obstructive Pulmonary Disease
Acronym: PH-6MST
Status: Completed | Type: Observational
Sponsor: ADIR Association (Other)
Responsible Party: Sponsor
Other Study IDs: PH-6MST
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Chronic Obstructive Pulmonary Disease; Pulmonary Rehabilitation; 6-minute Stepper Test
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective observational cohort: Every patient referred to pulmonary rehabilitation program will be eligible. They will perform cardiopulmonary exercise testing prior to join rehabilitation program.
  During the first session of pulmonary rehabilitation, they will perform 2 6-minute stepper test with a rest of 20 minutes minimum between each test.
  For the purpose of this study, patients will be offered to participate in an additional exercise session in which they will repeat the same procedure (two 6-minute stepper test) but but monitoring cardiopulmonary parameters and gaz exchanges using a face mask, a pneumotachograph and a gaz analyser (indirect calorimetry).
  Interventions: Other: 2 times : 6-minute stepper test with cardiorespiratory parameters and gaz exchange monitoring (with a rest of 20min between each test).

INTERVENTIONS:
Other: 2 times : 6-minute stepper test with cardiorespiratory parameters and gaz exchange monitoring (with a rest of 20min between each test). — For the 6-minute stepper test, please refer to NCT02842463 and NCT04004689. Gaz exchange analyzer will be calibrate before every test. Data will be recorded breath by breath.
  Heart rate will be monitored using a 12-lead electrocardiogram. Transcutaneous oxygen saturation will be assessed using a pulse oxymetry system at the earlobe.

SUMMARY:
Chronicle obstructive pulmonary disease is a worldwide cause of mortality and morbidity. This systemic disease progressively leads to dyspnea, muscle wasting and exercise capacity impairment.

Pulmonary rehabilitation is a cornerstone in the management of these systemic effects. Unfortunately, access to pulmonary rehabilitation is limited for many people who would benefit from it, primarily because of a lack of pulmonary rehabilitation and assessment centers. Optimal assessment should include an incremental cardiopulmonary exercise testing. This test allows to evaluate the factors contributing to exercise intolerance by linking performance and physiological parameters to the underlying metabolism. Moreover, it is the standard test to determine both the optimal training settings as well as any cardiopulmonary contraindications to pulmonary rehabilitation. However, this test is not available in most centers and when it is, consultations are limited. Therefore, pulmonary rehabilitation is often delayed for several weeks and patients can lose motivation.

In order to promote pulmonary rehabilitation, the incremental cardiopulmonary exercise testing could be replaced by field tests to individualize pulmonary rehabilitation prescription.

The six-minute stepper test is a new field tool. Its sensitivity and reproducibility have previously been reported in patients with chronicle obstructive pulmonary disease. It is easy to set up in the clinical setting and could be used to individualize pulmonary rehabilitation.

The main drawback when using field test is that they only provide a non specific assessement of the functional capacity because cardiopulmonary parameters and gaz exchanges are not monitored.

Although the performance during the 6-minute stepper test is moderately related with the maximal oxygen consumption during the incremental cardiopulmonary exercise testing performed on a cycloergometer, a direct comprehensive comparison of cardiopulmonary parameters and gaz exchanges during these two tests have never been performed.

Moreover, stepping is more closely related with activities of daily life (requiring a repetitive transition from rest to submaximal exercise intensity) than the maximal incremental exercise on cycloergometer and could provide further insight on the disability of patients during their usual activities, such as stair climbing (which is frequently avoided). Additionally, on-transient phase two oxygen consumption kinetic is particularly relevant because it evaluation is independent of the patient's motivation or criteria used to terminate exercise.

Therefore, the aim of this study is to compare the cardiorespiratory parameters, the gaz exchanges and the maximality between the six-minute stepper test and the incremental cardiopulmonary exercise testing performed on a cycloergometer.

The secondary objective was to compare the on-transient oxygen consumption phase two kinetic parameters (time constant, span and steady state) according to the severity of the disease.

DETAILED DESCRIPTION:
Experimental design:

This study is a pre-specified ancillary study to two other studies (with exactly the same design but a different population) aimed to assess the usability of the six-minute stepper test to prescribe endurance training in patients with mild to moderate (NCT02842463) and severe to very severe (NCT04004689) chronicle obstructive pulmonary disease respectively.

Patients already participating in one of these studies will be approached and offered to participate in an additional testing session (on a different day) using exactly the same procedure but monitoring cardiopulmonary parameters and gaz exchanges using a face mask, a pneumotachograph and a gaz analyser (indirect calorimetry).

Data from these additional two six-minute stepper tests will be compared with those obtained from the previously performed incremental cardiopulmonary exercise testing.

According to the American Thoracic Society and American College of Chest Physicians statement on cardiopulmonary exercise testing, maximality will be considered if either one or more of the following criteria occured:

1. The patient achieves predicted peak oxygen uptake and/or a plateau is observed.
2. Predicted maximal heart rate is achieved (>90%)
3. There is evidence of ventilatory limitation (breathing reserve <11liters or < 15%)
4. Respiratory exchange ratio > 1.15
5. Patient exhaustion/Borg Scale rating of 9-10 on a 0-to-10 scale.

Phase II oxygen consumption kinetics will be modelized by averaging the breath by breath measurement over consecutive periods of 5s for using the following monoexponential equation :

VO2 (τ) = VO2rest + VO2ss - VO2rest))*(1-e-t/τ). with " VO2rest " representing the baseline level of VO2 at rest, " VO2ss " representing the steady state of VO2 during exertion and τ (time constant) representing the time course of the monoexponential VO2 curve. The amplitude of the VO2 (VO2span) corresponds to the difference between VO2ss and VO2rest.

A curve by curve analysis will be performed across participants and parameters (time constant, span and steady state oxygen consumption) will be compared according to the stage of severity.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 ans ;
* Chronicle obstructive pulmonary disease stage I/IV ;
* Weight ≤ 90kg ;
* Eligible for pulmonary rehabilitation.

Exclusion Criteria:

* Require during exercise oxygen ;
* Pregnant woman or likely to be ;
* Patient under guardianship ;
* Contraindication to cardiopulmonary exercise testing ;
* Patient medically treated with heart rate modulator (excluding oral B2-agonist) ;
* Patient treated with pacemaker or defibrillator ;
* History of lower limb impairment (i.e. peripheral artery disease, orthopedic disorder etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronicle obstructive pulmonary disease reffered for pulmonary rehabilitation.
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Oxygen consumption using indirect calorimetry | The 2 6-minute stepper test will be carried out on the same day (20 minute of rest between each test) for a total time frame of 1 day.
  The tests will be performed using a face mask, a pneumotachograph and a gaz analyzer.

SECONDARY OUTCOMES:
Steps during 6-minute stepper test using stepper device. | The 2 6-minute stepper test will be carried out on the same day (20 minute of rest between each test) for a total time frame of 1 day.
Carbon dioxide production using indirect calorimetry | The 2 6-minute stepper test will be carried out on the same day (20 minute of rest between each test) for a total time frame of 1 day.
  The tests will be performed using a face mask, a pneumotachograph and a gaz analyzer.
Heart rate using a 12-lead electrocardiogram | The 2 6-minute stepper test will be carried out on the same day (20 minute of rest between each test) for a total time frame of 1 day.
  Heart rate wil be continuously monitored throughout the tests.
Transcutaneous oxygen saturation using a pulse oxymetry system | The 2 6-minute stepper test will be carried out on the same day (20 minute of rest between each test) for a total time frame of 1 day.
  Transcutaneous oxygen saturation will be continuously monitored throughout the tests at the earlobe.
Tidal volume using a pneumotachograph | The 2 6-minute stepper test will be carried out on the same day (20 minute of rest between each test) for a total time frame of 1 day.
  The outcome will be continuously monitored throughout the tests.
Respiratory rate using a pneumotachograph | The 2 6-minute stepper test will be carried out on the same day (20 minute of rest between each test) for a total time frame of 1 day.
  The outcome will be continuously monitored throughout the tests.
Minute ventilation using a pneumotachograph | The 2 6-minute stepper test will be carried out on the same day (20 minute of rest between each test) for a total time frame of 1 day.
  The outcome will be continuously monitored throughout the tests.
Respiratory exchange ratio using indirect calorimetry | The 2 6-minute stepper test will be carried out on the same day (20 minute of rest between each test) for a total time frame of 1 day.
  The outcome will be continuously monitored throughout the tests.
Oxygen equivalent using indirect calorimetry | The 2 6-minute stepper test will be carried out on the same day (20 minute of rest between each test) for a total time frame of 1 day.
  The outcome will be continuously monitored throughout the tests and calculated as the ratio between minute ventilation to oxygen consumption
Carbon dioxide equivalent using indirect calorimetry | The 2 6-minute stepper test will be carried out on the same day (20 minute of rest between each test) for a total time frame of 1 day.
  The outcome will be continuously monitored throughout the tests and calculated as the ratio between minute ventilation to carbon dioxide production
Ratio between dead space volume to tidal volume using a pneumotachograph and indirect calorimetry | The 2 6-minute stepper test will be carried out on the same day (20 minute of rest between each test) for a total time frame of 1 day.
  The outcome will be continuously monitored throughout the tests.
Dyspnea using the Borg scale | The 2 6-minute stepper test will be carried out on the same day (20 minute of rest between each test) for a total time frame of 1 day.
  Borg scale range from 0 (no breathlessness) to 10 (maximal breathlessness)
Lower limb fatigue using the Borg scale | The 2 6-minute stepper test will be carried out on the same day (20 minute of rest between each test) for a total time frame of 1 day.
  Borg scale range from 0 (no breathlessness) to 10 (maximal breathlessness)

CONTACTS AND LOCATIONS:
Overall Officials: David Debeaumont, MD, Principal Investigator — CHU-Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Service de physiologie urinaire, digestive, respiratoire et sportive, Bois-Guillaume, France; Catherine Tardif, MD, Study Chair — CHU-Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Service de physiologie urinaire, digestive, respiratoire et sportive, Bois-Guillaume, France; Antoine Cuvelier, Prof, PhD, Study Chair — CHU-Hôpitaux de Rouen - Service de pneumologie, Hôpital de Bois-Guillaume, Rouen, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France.; Tristan Bonnevie, MsC, Study Chair — ADIR Association, Bois-Guillaume, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France; Francis-Edouard Gravier, PT, Study Chair — ADIR Association, Bois-Guillaume, France; Catherine Viacroze, MD, Study Chair — CHU-Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Service de pneumologie, Bois-Guillaume, France; Jean-François Muir, Prof, PhD, Study Chair — CHU-Hôpitaux de Rouen - Service de pneumologie, Hôpital de Bois-Guillaume, Rouen, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France ; ADIR Association, Bois-Guillaume, France; Bouchra Lamia, Prof, PhD, Study Chair — UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France ; Service de pneumologie, Hôpital Jacques Monod 76290 Montivilliers; Jean Quieffin, MD, Study Chair — Service de pneumologie, Hôpital Jacques Monod 76290 Montivilliers; Guillaume Prieur, PT, MsC, Study Chair — Service de pneumologie, Hôpital Jacques Monod 76290 Montivilliers; Clément Médrinal, PT, MsC, Study Chair — UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France. Service de réanimation, Groupe Hospitalier du Havre, France; Pierre-Alexandre Hauss, MD, Study Chair — Service de pneumologie, Centre Hosptalier Intercommunal Elbeuf-Louviers-Val de Reuil
Locations (3):
- France (3):
  - ADIR Association, Bois-Guillaume
  - Centre Hostalier Intercommunal Elbeuf-Louviers-Val de Reuil, Elbeuf
  - Groupe Hospitalier du Havre, Le Havre